CLINICAL TRIAL: NCT06145529
Title: Resistance Training Based on Gamification During Physical Education
Brief Title: Resistance Training Based on Gamification in Children Aged 10-12 Years Old During Physical Education
Acronym: RETRAGAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: UV_INV_ETICA_2681359
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Muscular Fitness
Keywords: muscular strength; resistance training; children; gamification; physical education; school intervention

STUDY DESIGN:
Intervention Model Description: This randomized controlled trial (RCT) investigates the impact of resistance training (RT) with and without gamification on 300 children aged 10-12. Conducted in Valencia, Spain, six schools are randomly selected and assigned to three groups: EG1 (RT program), EG2 (RT with gamification), and CG (control). Participants are from grades 5 and 6, selected based on specific criteria. Interventions replace 15 minutes of PE in intervention schools. Sample size, determined for muscular fitness outcome, is ≃300 to account for potential dropout. Data analysis involves ANCOVA and multi-factor ANOVA, controlling for confounders. The study has received ethics approval.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EG1: 15 min RT (FunctionalHIIT) circuit program (Experimental): Volume: ≃10 min/day three times per week at moderate to high intensity (7-10 RPE). Intensity: During the study the children will instruct to follow the movements targeting firstly 6-7 and 9-10 at the end. Frequency: 3 times per week. Type of exercise: For the FunctionalHIIT program the participants will perform eight weight-bearing exercises in circuit format (i.e., push-ups, squats, planks, etc.). Training load variation: Initially, participants will start at an intensity level of 6-7 on the Borg's CR-10 scale, and this will increase by 1 point every two weeks until reaching 9-10 out of 10. The training duration during the main portion will increase by 5 seconds every two weeks, while the recovery interval between exercises will decrease. The exercises themselves will become progressively more challenging over the course of the training program and change every two weeks.
  Interventions: Other: RT Functional HIIT circuit program (15 minutes) with or without gamification approach
- EG2: 15 min RT (FunctionalHIIT) circuit program with gamification (Experimental): The EG2 training part will develop following the same protocol described in EG1.For the gamification experience, students will embark on a superhero-themed narrative journey where they must train diligently to earn points and badges, improving their avatars along the way. The ultimate goal is to defeat a super villain in the final battle after 8 weeks. The RETRAGAM study utilizes a self-created app (accessible at https://goo.su/GVgSPW) for the gamification story, point tracking, and personalization of children's avatars. As part of the flipped classroom approach, children can access the platform to preview upcoming exercises and educational content (i.e., benefits of RT, knowledge of the muscles, bones and joints involved in exercises, postural habits, etc.).
  Interventions: Other: RT Functional HIIT circuit program (15 minutes) with or without gamification approach
- CG (Control group) (No Intervention): We will provide general advice to the CG participants though an information meeting that will indicated to maintain their lifestyle. At the end of the intervention, in order to comply with the ethical commitment, PE teachers will be instructed on the RT programme and the RETRAGAM app to allow them to carry out the intervention autonomously when they consider.

INTERVENTIONS:
Other: RT Functional HIIT circuit program (15 minutes) with or without gamification approach — EG1 (RT Functional HIIT circuit program): This intervention involves a 15-minute Resistance Training (RT) Functional High-Intensity Interval Training (HIIT) circuit program. The focus is on functional movements performed at a high intensity within intervals.
  EG2 (RT Functional HIIT circuit program with gamification): This intervention replicates the RT Functional HIIT circuit program from EG1 but incorporates gamification strategies. Gamification involves the application of game-like elements, such as points, rewards, and competition, to make the exercise routine more engaging and enjoyable for the participants.
  Control Group (CG): Children in the control group continue with their regular Physical Education (PE) sessions, maintaining their usual routine
  Arms: EG1: 15 min RT (FunctionalHIIT) circuit program; EG2: 15 min RT (FunctionalHIIT) circuit program with gamification

SUMMARY:
For this investigation a total of ≃300 children (grades 5 and 6; 10-12 years of age) from 6 randomly selected schools in Valencia (Spain) will be enrolled during 8 weeks in one of the experimental groups (EG): EG1 (15' of RT Functional HIIT circuit program), EG2 (the same EG1 program but with a gamification approach) or CG (control group). Outcomes will include age and sex, maturity, PA profile, MF (assessed using an ad hoc battery), anthropometry and body composition (weight, height, sitting height, waist circumference and BMI) as well as the enjoyment and motivation during physical education. An interactive app in a digital device will be used for the gamification story, the point's registration with the personal children's avatar and content learning by flipped classroom. The hypothesis of the RETRAGAM study posits that children who participate in the gamified RT intervention will experience greater improvements in MF, body composition, motivation, and enjoyment compared to those who carry out the same intervention without gamification, as well as the control group (CG). Thus, the primary aim of the RETRAGAM study is to examine the effectiveness of a school-based RT intervention on MF, body composition, motivation, and enjoyment in children aged 10 to 12 years. Additionally, the study will compare the effects on the main outcomes among several intervention groups (i.e., RT, RT with gamification approach and the CG).

DETAILED DESCRIPTION:
Study design, participants and selection criteria The RETRAGAM study is a randomized controlled trial conducted in public primary schools in Valencia, Spain, with approval from The Human Research Ethics Committee of the Universitat of Valencia (Id: UV-INV_ETICA-2681359). The study aims to investigate the impact of a resistance training intervention with and without gamification on children aged 10-12 years.

To select the participating schools, random schools from a total of 167 primary schools in Valencia will be contacted by phone to inquire about their compliance with the inclusion criteria. Researchers will explain the study's main objectives, and once 6 schools meeting all the requirements are identified, they will be enrolled in the study. Each school will then be randomly assigned to one of three groups: EG1, EG2, or the CG. Within each school, one grade 5 and one grade 6 class will be randomly selected for the study. Subsequently, researchers will conduct a meeting with the school staff, to discuss the study's main objectives and the intervention procedure.

Among the three intervention schools selected, one will implement a 15-minute RT circuit program (EG1, n≃100), another will apply the same program but including gamification strategies (EG2, n≃100). The remaining school will serve as the control group (CG, n≃100). In the intervention schools, the first 15 minutes of PE lessons, typically allocated for warm-up, will be replaced by the RT circuit program. In the CG school, children will continue with their regular PE sessions.

To determine the sample size for the study, effect sizes for the primary outcome, muscular fitness, were estimated. While the health benefits of muscular fitness are widely acknowledged, there is a lack of consensus regarding the clinical significance of changes in MF in young people. Based on a prior study (Lubans et al., 2016), an effect size d=0.4 for MF is anticipated. Accordingly, a minimum sample of 162 children (54 per intervention group × 3 groups) is required to detect between-group changes in MF with a power of 80% and α=0.05. To account for potential dropout in a school context (up to 10%), the recruitment target is 145 children. However, to ensure an ample number of participants, ≃300 students will be recruited (≃100 per intervention group).

Interventions

Considering that school-based RT interventions should be realistic, adapted to the school timetable, and focused on improve MF, body composition, enjoyment and motivation in primary school children 10-12 years aged, the following four 8-week school-based interventions programs were chosen for this study:

The two-interventions included in the RETRAGAM study have been designed by the researcher based on suggestions regarding the desirability of exercises to specifically develop MF following the RT guidelines for children and adolescents (Faigenbaum et al., 2009b; Lloyd et al., 2014) and considering previous developed interventions in the same range of age (Villa-González et al., 2022).

EG1: 15 min RT (FunctionalHIIT) circuit program High intensity interval training (HIIT) describes physical exercise characterized by short and intermittent efforts of vigorous activity, interspersed with resting periods at passive or low-intensity exercises (Amaro-Gahete et al., 2018). During each FunctionalHIIT training the teacher will demonstrate performance movements and will give feedback to students considering the correct execution providing standardized verbal encouragement.

Volume: ≃10 min/day three times per week at moderate to high intensity (7-10 in the Borg's CR-10 scale) (Borg, 1990) a total of ≃30 min/week, which will be the half than the minimum children's PA recommended by the WHO (60 min/week at MVPA).

Intensity: Participants were familiarized with the Borg's CR-10 scale (Borg, 1990) before the start of the intervention. During the study the children will instruct to follow the movements targeting firstly 6-7 and 9-10 at the end. After each FunctionalHIIT training, all students will rate their perceived exertion during exercise. Although there are previous studies that control intensity using the Borg scale in children of these ages (Chen et al., 2017; Engel et al., 2019; Moran et al., 2019), some random students belong to all groups (i.e., EG1, EG2 and CG) will wear a heart rate monitor (Polar Ignite 2 monitor) to control different intensity parameters (i.e., HR, HRMax, HRV).

Frequency: 3 times per week, based on a previous intervention on FunctionalHIIT in children (Engel et al., 2019) and following the RT guidelines for children and adolescents (Faigenbaum et al., 2009b; Stricker et al., 2020) and the recommendations of the Resistance Training for Children Consensus (Lloyd et al., 2014).

Type of exercise: For the FunctionalHIIT program the participants will perform eight weight-bearing exercises in circuit format (i.e., push-ups, squats, planks, etc.).

Training load variation: We consider that participants will not immediately meet the required intensity level. Instead, a gradual progression will be introduced to control the exercise dose. Initially, participants will start at an intensity level of 6-7 on the Borg's CR-10 scale, and this will increase by 1 point every two weeks until reaching 9-10 out of 10. The training duration during the main portion will increase by 5 seconds every two weeks, while the recovery interval between exercises will decrease (from 3 seconds initially to 15 seconds at the end). The exercises themselves will become progressively more challenging over the course of the training program and change every two weeks. Furthermore, considering individual characteristics, the progression will be adapted for particularly inactive or overweight children, allowing them to repeat exercises from the previous week.

Training sessions: Each training session will commence with a 3-minute dynamic standardized warm-up (3-6 RPE), including muscle activation exercises such as skipping, jumping jacks, and jumps. The 10-minute main part (7-10 RPE) will involve participants performing eight exercises in pairs or trios in a circuit format, with a focus on making as many repetitions as possible and targeting the previously indicated RPE levels. The teacher, along with the support of two selected students from the school, will encourage and monitor the technique and effort during the circuit. The training session will conclude with a 2-minute cooling-down (3-4 RPE) that includes stretching exercises.

EG2: 15 min RT (FunctionalHIIT) circuit program with gamification The EG2 training part will develop following the same protocol described in EG1.For the gamification experience, students will embark on a superhero-themed narrative journey where they must train diligently to earn points and badges, improving their avatars along the way. The ultimate goal is to defeat a super villain in the final battle after 8 weeks. The RETRAGAM study utilizes a self-created app (accessible at https://goo.su/GVgSPW) for the gamification story, point tracking, and personalization of children's avatars. As part of the flipped classroom approach, children can access the platform to preview upcoming exercises and educational content (i.e., benefits of RT, knowledge of the muscles, bones and joints involved in exercises, postural habits, etc.). To motivate students, biweekly motivational videos related to the superhero narrative will be shared, encouraging them to actively participate in the RT program. At the end of each training day, students will conduct self-evaluations, earning 0-3 points based on their level of training engagement (exercise technique, RPE compliance and comradeship). These points will be used to improve their individual avatars at the end of each week (i.e., superhero attires, equipment, power, etc.). At the end of the 8 weeks, students will have to defeat the super villain at the final battle (questionnaire on what has been learned) and they will receive a physical badge that they can wear in their t-shirt at the retest measurement session. Teacher will have a spreadsheet to record all the points that will complement the evaluation of the PE sessions. Figure 1 summarises the EG2 intervention.

CG (Control group) We will provide general advice to the CG participants though an information meeting that will indicated to maintain their lifestyle. At the end of the intervention, in order to comply with the ethical commitment, PE teachers will be instructed on the RT programme and the RETRAGAM app to allow them to carry out the intervention autonomously when they consider.

Data analysis All outcome variables will be verified for normality, and the results will be presented using mean and standard deviation or median and interquartile range, where appropriate for continuous variables, and frequency and percentage for categorical variables. We will use an analysis of covariance (ANCOVA) for between group comparisons at the baseline (EG1 vs EG2 vs CG), and the nonparametric method of Kruskal-Wallis and t-tests, as appropriate.

To assess the effectiveness of the different interventions on objectively measured MF and the other outcomes, a multi-factor ANOVA [time-point (T0, T1) x group (EG1 vs EG2 vs CG)] will be used with the outcome measures as dependent variables in separate models, the intervention as an independent variable and controlling for potential confounders (such as gender, sociodemographic characteristics, health status, BMI, PHV, PA level and MF baseline). Statistical significance will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

As this is a school-based intervention study, the inclusion criteria are for the school itself. They are as follows:

1. 1 class of grade 5 and other of grade 6 in the school.
2. At least 20 children class size.
3. Includes 45 min PE sessions three times per week in both grades.
4. They cannot develop physical condition didactic unite at the same time.

Exclusion Criteria:

* Exclusion criteria include participants who have diagnosed medical problems that prevent them from participating in the intervention.

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-05 (Estimated)

PRIMARY OUTCOMES:
Muscular fitness (MF) | this outcome will be assessed twice: a pre-test two weeks before the 8-week intervention and a post-test one week after the intervention.
  MF will be assessed using a battery of children strength designed ad hoc for this investigation. This battery comprises 8 tests that assess the 3 dimensions of MF: strength, power, and endurance. These tests encompass upper limbs (handgrip, push-up test, and medicinal ball throwing), lower limbs (single-hop test, two-legged squat test, and standing long jump), and trunk strength (curl-up test and sport-specific endurance plank test). Before the fitness assessments, all participants will engage in a 5-minute dynamic standardized warm-up, involving exercises that activate the muscles and improve joint mobility, such as limb mobility exercises, skipping, jumping jacks, and jumps.

SECONDARY OUTCOMES:
Sociodemographic characteristics and health status | this outcome will be assessed twice: a pre-test two weeks before the 8-week intervention and a post-test one week after the intervention.
  Families will complete a questionnaire about the child's sociodemographic characteristics including date of birth and gender, household factors, family's socioeconomic status (family income, parental education, and parental employment status), and the child's health status (reporting medical conditions and medications, if any)
Anthropometric Data and Body Composition | this outcome will be assessed twice: a pre-test two weeks before the 8-week intervention and a post-test one week after the intervention.
  Anthropometric assessments will be conducted on participants following International Standards for Anthropometric Assessment (ISAK). Weight, height, sitting height, and waist circumference will be measured using specific protocols. Weight, assessed with a Tanita BC-601 system, will be checked for zero reading before participants stand evenly on the scales. Height, measured with a Seca stadiometer, will follow the stretch stature method. Sitting height, also measured with the Seca stadiometer, involves a seated position on a known-height chair. Waist circumference, measured with a Seca 201 tape, is taken at the narrowest point between the lower costal border and the iliac crest. Neck circumference is measured similarly, immediately superior to the thyroid cartilage. Each measurement will be taken twice, and the average used in analysis. Body mass index (BMI) will be calculated as weight in kilograms divided by the square of height in meters.
Maturity | this outcome will be assessed twice: a pre-test two weeks before the 8-week intervention and a post-test one week after the intervention.
  Peak Height Velocity (PHV), a somatic biological maturity indicator, signifies the maximum growth velocity during adolescence. Determined by gender, date of birth, height, sitting height, and weight, it is calculated using gender-specific multiple-regression equations available on the SCGD research group website. The website predicts an individual's proximity to PHV (years from age at PHV). Designed for ages 8-16 in females and 9-18 in males, with a maturity age range of -4 to +4 years from PHV. Categorization includes Pre-PHV (before puberty), Circa-PHV (during puberty), and Post-PHV (after puberty), using specific value ranges. To avoid biases, values between 0.5-1 and -1 to -0.5 are considered missing data in this study.
Physical Activity Profile | this outcome will be assessed twice: a pre-test two weeks before the 8-week intervention and a post-test one week after the intervention.
  Physical activity (PA) assessment in the study will use the Youth Activity Profile (YAP), a subjective tool developed to evaluate PA and sedentary habits in children and adolescents. The YAP-S, a Spanish adaptation, was created as an alternative to objective PA measurements using accelerometers or pedometers. It consists of 19 questions, covering general engagement and enjoyment of PA, as well as specific PA and sedentary habits over the previous week. The questionnaire is translated and adapted by the PROFITH group and is considered a feasible and reliable tool for assessing PA and sedentary behavior in Spanish children and adolescents. The information collected is categorized into "Physical activity at school," "Physical activity outside school," and "Sedentary habits" based on the context in which it was developed.
Enjoyment and motivation | this outcome will be assessed twice: a pre-test two weeks before the 8-week intervention and a post-test one week after the intervention.
  The RETRAGAM study will assess enjoyment and motivation during physical education (PE) using two scales: the Physical Activity Enjoyment Scale (PACES) and the Situational Motivation Scale in PE. The Spanish version of PACES, consisting of 16 items, gauges enjoyment levels during physical activity, ranging from the highest to lowest. Responses, on a Likert scale from 1 to 5, reflect agreement or disagreement. The Situational Motivation Scale in PE, with 16 items, measures motivation factors in PE activities, categorized into intrinsic motivation, identified regulation, external regulation, and demotivation. Participants rate each item on a 7-point Likert scale, indicating their level of agreement. Both scales provide valuable insights into enjoyment and motivation levels during PE lessons in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Molina-García, Study Director — University of Valencia
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amaro-Gahete FJ, De-la-O A, Jurado-Fasoli L, Espuch-Oliver A, Robles-Gonzalez L, Navarro-Lomas G, de Haro T, Femia P, Castillo MJ, Gutierrez A. Exercise training as S-Klotho protein stimulator in sedentary healthy adults: Rationale, design, and methodology. Contemp Clin Trials Commun. 2018 May 18;11:10-19. doi: 10.1016/j.conctc.2018.05.013. eCollection 2018 Sep. PMID 30023455
- [Background] Borg G. Psychophysical scaling with applications in physical work and the perception of exertion. Scand J Work Environ Health. 1990;16 Suppl 1:55-8. doi: 10.5271/sjweh.1815. PMID 2345867
- [Background] Buchan DS, Young JD, Simpson AD, Thomas NE, Cooper SM, Baker JS. The effects of a novel high intensity exercise intervention on established markers of cardiovascular disease and health in Scottish adolescent youth. J Public Health Res. 2012 May 25;1(2):155-7. doi: 10.4081/jphr.2012.e24. eCollection 2012 Jun 15. PMID 25170459
- [Background] Bull FC, Al-Ansari SS, Biddle S, Borodulin K, Buman MP, Cardon G, Carty C, Chaput JP, Chastin S, Chou R, Dempsey PC, DiPietro L, Ekelund U, Firth J, Friedenreich CM, Garcia L, Gichu M, Jago R, Katzmarzyk PT, Lambert E, Leitzmann M, Milton K, Ortega FB, Ranasinghe C, Stamatakis E, Tiedemann A, Troiano RP, van der Ploeg HP, Wari V, Willumsen JF. World Health Organization 2020 guidelines on physical activity and sedentary behaviour. Br J Sports Med. 2020 Dec;54(24):1451-1462. doi: 10.1136/bjsports-2020-102955. PMID 33239350
- [Background] Burgueño, R., Granero-Gallegos, A., Alcaráz-Ibáñez, M., Sicilia, A., Medina-Cusabón, J. (2018). La necesidad de medir la motivación situacional en el contexto español de la educación física: Psicometría de la Situational Motivation Scale. Cuadernos de Psicología del Deporte, 18(2), 135-151
- [Background] Chen YL, Chiou WK, Tzeng YT, Lu CY, Chen SC. A rating of perceived exertion scale using facial expressions for conveying exercise intensity for children and young adults. J Sci Med Sport. 2017 Jan;20(1):66-69. doi: 10.1016/j.jsams.2016.05.009. Epub 2016 Jun 1. PMID 27267301
- [Background] Chillon P, Galvez-Fernandez P, Huertas-Delgado FJ, Herrador-Colmenero M, Barranco-Ruiz Y, Villa-Gonzalez E, Aranda-Balboa MJ, Saucedo-Araujo RG, Campos-Garzon P, Molina-Soberanes D, Segura-Diaz JM, Rodriguez-Rodriguez F, Lara-Sanchez AJ, Queralt A, Molina-Garcia J, Bengoechea EG, Mandic S. A School-Based Randomized Controlled Trial to Promote Cycling to School in Adolescents: The PACO Study. Int J Environ Res Public Health. 2021 Feb 20;18(4):2066. doi: 10.3390/ijerph18042066. PMID 33672550
- [Background] Eken MM, Harlaar J, Dallmeijer AJ, de Waard E, van Bennekom CA, Houdijk H. Squat test performance and execution in children with and without cerebral palsy. Clin Biomech (Bristol). 2017 Jan;41:98-105. doi: 10.1016/j.clinbiomech.2016.12.006. Epub 2016 Dec 18. PMID 28040656
- [Background] Engel FA, Wagner MO, Schelhorn F, Deubert F, Leutzsch S, Stolz A, Sperlich B. Classroom-Based Micro-Sessions of Functional High-Intensity Circuit Training Enhances Functional Strength but Not Cardiorespiratory Fitness in School Children-A Feasibility Study. Front Public Health. 2019 Nov 14;7:291. doi: 10.3389/fpubh.2019.00291. eCollection 2019. PMID 31799229
- [Background] Eurofit (1993). Handbook for the EUROFIT tests of Physical Fitness. 2nd ed. Strasbourg: Council of Europe, Commitee for the Development of Sport. 75 p.
- [Background] Faigenbaum AD, Kraemer WJ, Blimkie CJ, Jeffreys I, Micheli LJ, Nitka M, Rowland TW. Youth resistance training: updated position statement paper from the national strength and conditioning association. J Strength Cond Res. 2009 Aug;23(5 Suppl):S60-79. doi: 10.1519/JSC.0b013e31819df407. PMID 19620931
- [Background] Faigenbaum AD, Bush JA, McLoone RP, Kreckel MC, Farrell A, Ratamess NA, Kang J. Benefits of Strength and Skill-based Training During Primary School Physical Education. J Strength Cond Res. 2015 May;29(5):1255-62. doi: 10.1519/JSC.0000000000000812. PMID 25536540
- [Background] Guay, F., Vallerand, R. J., & Blanchard, C. (2000). On the assessment of situational intrinsic and extrinsic motivation: The Situational Motivation Scale (SIMS). Motivation and emotion, 24(3), 175-213. doi:10.1023/A:1005614228250
- [Background] Lloyd RS, Faigenbaum AD, Stone MH, Oliver JL, Jeffreys I, Moody JA, Brewer C, Pierce KC, McCambridge TM, Howard R, Herrington L, Hainline B, Micheli LJ, Jaques R, Kraemer WJ, McBride MG, Best TM, Chu DA, Alvar BA, Myer GD. Position statement on youth resistance training: the 2014 International Consensus. Br J Sports Med. 2014 Apr;48(7):498-505. doi: 10.1136/bjsports-2013-092952. Epub 2013 Sep 20. PMID 24055781
- [Background] Lubans DR, Smith JJ, Peralta LR, Plotnikoff RC, Okely AD, Salmon J, Eather N, Dewar DL, Kennedy S, Lonsdale C, Hilland TA, Estabrooks P, Finn TL, Pollock E, Morgan PJ. A school-based intervention incorporating smartphone technology to improve health-related fitness among adolescents: rationale and study protocol for the NEAT and ATLAS 2.0 cluster randomised controlled trial and dissemination study. BMJ Open. 2016 Jun 27;6(6):e010448. doi: 10.1136/bmjopen-2015-010448. PMID 27354070
- [Background] Marfell-Jones, M. J., Stewart, A. D., & De Ridder, J. H. (2012). International standards for anthropometric assessment.
- [Background] Martínez, E. (2002). Pruebas de aptitud física. España, Barcelona: Paidotribo.
- [Background] Moran CA, Corso SD, Bombig MT, Serra AJ, Pereira SA, Peccin MS. Heart rate agreement between the 20-meter shuttle run test and virtual system in healthy children: a cross-sectional study. BMC Pediatr. 2019 Dec 12;19(1):491. doi: 10.1186/s12887-019-1861-4. PMID 31830948
- [Background] Moreno, J. A., González-Cutre, D., Martínez, C., Alonso, N., & López, M. (2008). Propiedades psicométricas de la Physical Activity Enjoyment Scale (PACES) en el contexto español. Estudios de Psicología, 29(2), 173-180. doi: 10.1174/021093908784485093
- [Background] Plowman, S.A. (2013). Muscular Strength, Endurance, and Flexibility Assessments. In S. A. Plowman & M.D. Meredith (Eds.), Fitnessgram/Activitygram Reference Guide (4th Edition) (pp. Internet Resource). Dallas, TX: The Cooper Institute, 8-1 - 8-55.
- [Background] Ruiz JR, Espana Romero V, Castro Pinero J, Artero EG, Ortega FB, Cuenca Garcia M, Jimenez Pavon D, Chillon P, Girela Rejon MJ, Mora J, Gutierrez A, Suni J, Sjostrom M, Castillo MJ. [ALPHA-fitness test battery: health-related field-based fitness tests assessment in children and adolescents]. Nutr Hosp. 2011 Nov-Dec;26(6):1210-4. doi: 10.1590/S0212-16112011000600003. Spanish. PMID 22411362
- [Background] Stricker PR, Faigenbaum AD, McCambridge TM; COUNCIL ON SPORTS MEDICINE AND FITNESS. Resistance Training for Children and Adolescents. Pediatrics. 2020 Jun;145(6):e20201011. doi: 10.1542/peds.2020-1011. PMID 32457216
- [Background] Tercedor P, Villa-Gonzalez E, Avila-Garcia M, Diaz-Piedra C, Martinez-Baena A, Soriano-Maldonado A, Perez-Lopez IJ, Garcia-Rodriguez I, Mandic S, Palomares-Cuadros J, Segura-Jimenez V, Huertas-Delgado FJ. A school-based physical activity promotion intervention in children: rationale and study protocol for the PREVIENE Project. BMC Public Health. 2017 Sep 26;17(1):748. doi: 10.1186/s12889-017-4788-4. PMID 28950837
- [Background] Tong TK, Wu S, Nie J. Sport-specific endurance plank test for evaluation of global core muscle function. Phys Ther Sport. 2014 Feb;15(1):58-63. doi: 10.1016/j.ptsp.2013.03.003. Epub 2013 Jul 11. PMID 23850461
- [Background] Villa-Gonzalez E, Barranco-Ruiz Y, Garcia-Hermoso A, Faigenbaum AD. Efficacy of school-based interventions for improving muscular fitness outcomes in children: A systematic review and meta-analysis. Eur J Sport Sci. 2023 Mar;23(3):444-459. doi: 10.1080/17461391.2022.2029578. Epub 2022 Apr 12. PMID 35023448